CLINICAL TRIAL: NCT00044785
Title: A Phase I Study of Escalating Doses of CPT-11 and 5fluorouracil (5FU) Plus PN401 With a Fixed Dose of Leucovorin in Patients With Solid Tumor Malignancies.
Brief Title: Phase I Study of PN401, Fluorouracil, Leucovorin and CPT-11 in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Wellstat Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 401.02.001; GCC0121
Record Dates: First submitted 2002-09-04; First posted 2002-09-06 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-05

CONDITIONS: Solid Tumors
Keywords: colorectal cancer; gastric cancer; breast cancer
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Breast Neoplasms | interventions — uridine triacetate; Fluorouracil; Leucovorin; Irinotecan

INTERVENTIONS:
Drug: triacetyluridine
Drug: fluorouracil
Drug: leucovorin
Drug: camptosar

SUMMARY:
CPT-11 and 5Fluorouracil (5FU) combined with leucovorin has become the standard of care for colorectal cancer. PN401 permits treatment with higher than normal doses of 5FU, which could increase its therapeutic potential. It is hypothesized that adding PN401 to the CPT-11, 5FU, leucovorin regimen will reduce toxicity and will allow higher doses of 5FU to be well tolerated and therefore potentially increase effectiveness.

ELIGIBILITY:
Inclusion Criteria

* Must be at least 18 years of age;
* Life expectancy: At least 3 months;
* Performance status: ECOG of 0 or 1;
* Histologic or cytologic proof of a solid tumor cancer that is not amenable to curative surgical resection;
* Evaluable or measurable disease documented within 4 weeks of the start of treatment;
* Prior chemotherapy or radiotherapy is allowed if 4 weeks or more have elapsed prior to starting treatment and patients have recovered from toxicities of prior treatment;
* Adequate organ function:

Hematopoietic: ANC = 1500/ul or more, Platelets = 100,000/ul or more, Hemoglobin = 9.5 g/dL or more, transfusion prior to evaluation is allowed; Hepatic: Bilirubin = 2.0 mg/dL or less and SGPT(ALT) and SGOT(AST) < 3 x upper limit of normal (< 5 x upper limit of normal if liver metastases present) Renal: Serum Creatinine < 2.0 mg/dL;

* Patient has the initiative, geographic proximity, and means to be compliant with the protocol;
* Fertile patients (male or female) must agree to use effective contraception;
* Must be able to swallow and retain tablets.

Exclusion Criteria

* Major surgery within the four weeks preceding the start of treatment;
* Serious medical or psychiatric illness that would prevent self-determined informed consent;
* Intensive chemotherapy treatment;
* Infection or antibiotics at the time of screening;
* Uncontrolled cardiovascular, pulmonary, renal, neurologic, psychiatric, or hepatic dysfunction;
* Pregnant or nursing;
* Pre-existing diarrhea or uncontrolled clinically significant illness other than cancer (i.e. ulcerative colitis, malabsorption syndrome);
* Brain metastases that have not been stable for more than 3 months;
* Known Dihydropyrimidine Dehydrogenase (DPD) deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2002-08; Study Completion 2004-03

PRIMARY OUTCOMES:
Safety and Maximum Tolerated Dose

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland, United States